CLINICAL TRIAL: NCT04910321
Title: Hangzhou Hospital Staff Cohort
Acronym: HHSC
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated due to the COVID-19 situation.
Sponsor: Westlake University (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Hangzhou Women's Hospital (Unknown); Red Cross Hospital, Hangzhou, China (Other)
Responsible Party: Sponsor
Other Study IDs: 20201221ZJS001
Record Dates: First submitted 2021-04-05; First posted 2021-06-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Metabolic Syndrome | interventions — Diet; Exercise; Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: diet, physical activities, sleep — lifestyle factors

SUMMARY:
The Hangzhou Hospital Staff Cohort (HHSC) is a prospective cohort study among staffs from three hospitals located in Hangzhou, China, including the Hangzhou First People's Hospital, Hangzhou Women's Hospital, and Hangzhou Red Cross Hospital. Participants recruitment and baseline survey including anthropometric, lifestyle and clinical measurement, as well as biological samples collection are initiated in January 2021. Recruited hospital staff are followed up every year during the medical examination organized by their employer. The primary aim of the HHSC study is to investigate the prospective associations of diet, physical activities, sleep, and other lifestyle factors with the long-term metabolic health of the hospital staffs. The secondary aim of the HHSC study is to integrate multi-omics data including genomics, metabolomics, proteomics and microbiome by a machine learning algorithm, to probe into the complex mediating roles of gene, metabolism and gut microbiota linking lifestyle factors with metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older
* Serving staffs of designated hospitals

Exclusion Criteria:

* Participants with cancer
* Participants with other serious medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are serving staffs from the Hangzhou Frirst People's Hospital, Hangzhou Women's Hospital, and Hangzhou Red Cross Hospital are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes diagnosed as fasting blood glucose larger than 7.0 mmol/L | 3 years after enrollment
  Fasting blood glucose is measured every year during follow-up
Incidence of type 2 diabetes diagnosed as fasting blood glucose larger than 7.0 mmol/L | 6 years after enrollment
  Fasting blood glucose is measured every year during follow-up
Incidence of type 2 diabetes diagnosed as fasting blood glucose larger than 7.0 mmol/L | 9 years after enrollment
  Fasting blood glucose is measured every year during follow-up

SECONDARY OUTCOMES:
Change of body mass index | Change from baseline at 3 years
  Participants' body weight and height was measured to calculate body mass index every year during follow-up
Change of body mass index | Change from baseline at 6 years
  Participants' body weight and height was measured to calculate body mass index every year during follow-up
Change of body mass index | Change from baseline at 9 years
  Participants' body weight and height was measured to calculate body mass index every year during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided